CLINICAL TRIAL: NCT00046267
Title: A Pilot Study of the Safety, Efficacy, and Tolerability of Extended-Release Niacin (Niaspan) for the Treatment of Elevated Non-HDL Cholesterol and Elevated Triglycerides in HIV-Infected Subjects
Brief Title: Niacin for Treatment of Elevated Cholesterol and Triglycerides in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5148
Record Dates: First submitted 2002-09-24; First posted 2002-09-25 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections; Hypercholesterolemia; Hypertriglyceridemia; Diabetes Mellitus
Keywords: Delayed-Action Preparations; Blood Glucose; Insulin; Alanine Transaminase; Aspartate Aminotransferases; Fructosamine; Glucose Tolerance Test; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hypercholesterolemia; Hypertriglyceridemia; Diabetes Mellitus; Insulin Resistance | interventions — Niacin

INTERVENTIONS:
Drug: Niacin

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and tolerability of extended-release niacin (Niaspan) in improving the level of fats in the blood of HIV-infected patients.

DETAILED DESCRIPTION:
Lipid disorders are common among patients with HIV and tend to worsen with potent antiretroviral therapy. Lipid-lowering drugs are not always effective, and few data address interactions between antiretroviral drugs and lipid-lowering agents. Additional agents for the treatment of lipid metabolism disorders in HIV-infected patients are needed. Niacin, which is highly effective for similar lipid disorders in the general population, may be effective in treating lipid disorders in patients with HIV.

This 48-week study consists of two steps. In Step 1, patients will begin a lipid-lowering diet and exercise regimen that will continue throughout the study. After 4 weeks on the regimen, patients will enter Step 2 of the study and will begin extended-release niacin therapy. During Step 2, niacin will be dose-escalated every 4 to 6 weeks over a 16-week period. At Weeks 14 and 20, the niacin dose will be determined by blood fat levels. Patients will remain on the dose set at Week 20 for the remainder for the study. If blood tests taken at Week 24 show that blood fat levels have not improved significantly, patients have the option of adding another fat-lowering drug to their therapy.

Patients will visit the clinic at entry and at Weeks 4, 8, 12, 18, 24, 32, 40, and 48. Patients may be asked to come to the clinic at Weeks 14 and 20 to receive additional study drug. Patients must fast for 8 to 12 hours before the screening visit and before each study visit in which blood will be drawn. Blood will be drawn throughout the study for fat, sugar, and insulin tests and for CD4 and CD8 cell counts.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected.
* Stable antiretroviral therapy for 3 months to 1 month prior to study entry and planning to stay on current therapy. No changes in antiretroviral therapy will be allowed in the 1-month period prior to study entry.
* Fasting non-HDL-C >= 180 mg/dl and serum triglycerides > 200 mg/dl within 30 days of study entry.
* Willing to stay on the Lipid-Lowering Diet and Activity Guide for the length of the study.
* Women of reproductive potential must have a negative serum or urine pregnancy test performed within 14 days prior to study entry.
* Agrees to use acceptable methods of contraception while receiving protocol-specified medication and for 4 weeks after stopping the medication. Patients who are not of reproductive potential are eligible without requiring the use of contraception.
* Men who have been on stable testosterone replacement for at least 3 months prior to entry and plan to continue a stable dose during the study may enroll.
* Hormone replacement therapy for postmenopausal women and for transgendered patients will be allowed, but not required. Oral contraceptive therapy will be allowed. Patients must be on stable hormone replacement therapy for at least 30 days prior to study entry and plan to continue a stable dose during the study.

Exclusion Criteria:

* LDL-C >= 200 mg/dl or non-HDL-C > 250 mg/dl (if the LDL-C cannot be calculated because the triglycerides are > 400 mg/dl).
* Coronary heart disease (CHD) or CHD risk equivalent, including but not limited to peripheral vascular disease, cerebrovascular disease, or abdominal aortic aneurysm.
* Congestive heart failure.
* Uncontrolled hypertension within 30 days of study entry, from an average of 2 or more readings on 2 or more occasions.
* Acute arthritic gout symptoms within 60 days of study entry.
* Active peptic ulcer disease.
* Diabetes mellitus that requires pharmacological or dietary control.
* Untreated hypothyroidism. Patients with treated hypothyroidism are allowed.
* Levothyroxine and liothyronine for uses other than for hypothyroidism.
* Active or symptomatic gallbladder disease within 1 year of study entry. Patients with asymptomatic gallstones are allowed. Patients with a history of a cholecystectomy will be allowed provided that the procedure was done at least 3 months before study entry.
* Active cancer within the last 5 years or a new diagnosis of cancer within the last 5 years. Skin cancers, including Kaposi's sarcoma, not requiring systemic treatment are allowed.
* Pregnancy or breast-feeding.
* Any prescription lipid-lowering agent within 30 days of study entry.
* Niacin or niacin-containing products that contain > 100 mg daily within 30 days prior to study entry.
* Systemic cancer chemotherapy or immunomodulators within 60 days of study entry.
* Investigational antiretroviral drugs in AACTG studies and expanded access trials will be allowed. Other investigational therapies that are not FDA-approved will not be allowed within 30 days of study entry unless permission is granted by study chairs.
* Systemic glucocorticoids above replacement levels within 60 days of entry.
* Certain antidiabetic medications.
* Allergy/sensitivity to the study drug or its formulations.
* Allergy, sensitivity, or severe intolerance to all of the following 3 medications: aspirin, ibuprofen, and naproxen.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Decreased mental capacity that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Active AIDS-defining opportunistic infection (OI) within 30 days prior to entry. Patients who have no evidence of active disease and are receiving maintenance therapy for AIDS-related OIs will be eligible.
* Acute illness within 30 days prior to entry that, in the opinion of the site investigator, would interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Dube, M. D., Study Chair; James H. Stein, M. D., Study Chair
Locations (16):
- United States (16):
  - UCLA School of Medicine, Los Angeles, California
  - Univ of California, San Diego Antirviral Research, San Diego, California
  - San Mateo County AIDS Program, Stanford, California
  - Stanford Univ, Stanford, California
  - Willow Clinic, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Indiana University Hospital, Indianapolis, Indiana
  - Methodist Hosp of Indiana, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - Univ of Minnesota, Minneapolis, Minnesota
  - St. Louis Connect Care, St Louis, Missouri
  - Washington Univ (St. Louis), St Louis, Missouri
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Dube MP, Sprecher D, Henry WK, Aberg JA, Torriani FJ, Hodis HN, Schouten J, Levin J, Myers G, Zackin R, Nevin T, Currier JS; Adult AIDS Clinical Trial Group Cardiovascular Disease Focus Group. Preliminary guidelines for the evaluation and management of dyslipidemia in adults infected with human immunodeficiency virus and receiving antiretroviral therapy: Recommendations of the Adult AIDS Clinical Trial Group Cardiovascular Disease Focus Group. Clin Infect Dis. 2000 Nov;31(5):1216-24. doi: 10.1086/317429. Epub 2000 Nov 7. PMID 11073755
- [Background] Mulligan K, Grunfeld C, Tai VW, Algren H, Pang M, Chernoff DN, Lo JC, Schambelan M. Hyperlipidemia and insulin resistance are induced by protease inhibitors independent of changes in body composition in patients with HIV infection. J Acquir Immune Defic Syndr. 2000 Jan 1;23(1):35-43. doi: 10.1097/00126334-200001010-00005. PMID 10708054
- [Background] McKenney JM, Proctor JD, Harris S, Chinchili VM. A comparison of the efficacy and toxic effects of sustained- vs immediate-release niacin in hypercholesterolemic patients. JAMA. 1994 Mar 2;271(9):672-7. PMID 8309029
- [Background] Guyton JR, Goldberg AC, Kreisberg RA, Sprecher DL, Superko HR, O'Connor CM. Effectiveness of once-nightly dosing of extended-release niacin alone and in combination for hypercholesterolemia. Am J Cardiol. 1998 Sep 15;82(6):737-43. doi: 10.1016/s0002-9149(98)00448-2. PMID 9761083
- [Background] Hadigan C, Meigs JB, Corcoran C, Rietschel P, Piecuch S, Basgoz N, Davis B, Sax P, Stanley T, Wilson PW, D'Agostino RB, Grinspoon S. Metabolic abnormalities and cardiovascular disease risk factors in adults with human immunodeficiency virus infection and lipodystrophy. Clin Infect Dis. 2001 Jan;32(1):130-9. doi: 10.1086/317541. Epub 2000 Dec 15. PMID 11118392